CLINICAL TRIAL: NCT06425302
Title: A Phase 2 Randomized, Open Label Study to Evaluate the Efficacy and Safety of Golcadomide in Combination With Rituximab in Participants With Newly Diagnosed Advanced Stage Follicular Lymphoma
Brief Title: A Study to Evaluate the Efficacy and Safety of Golcadomide in Combination With Rituximab in Participants With Newly Diagnosed Advanced Stage Follicular Lymphoma
Acronym: GOLSEEK-2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA073-1022; U1111-1303-4594 (Other: WHO); 2024-511304-16 (Other: EU CTR)
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma, Follicular
Keywords: Follicular lymphoma; Grade 1-3a Follicular lymphoma; BMS-986369; CC-99282; Lymphoma; golcadomide
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma | interventions — Rituximab; Cyclophosphamide; Doxorubicin; liposomal doxorubicin; 1-dodecylpyridoxal; Vincristine; Prednisone; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Rituximab + Chemotherapy (Experimental): R-CHOP (Rituximab, Doxorubicin, Vincristine, Cyclophosphamide, Prednisone) or Rituximab + Bendamustine
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Bendamustine
- Golcadomide Dose 1 + Rituximab (Experimental)
  Interventions: Drug: Golcadomide; Drug: Rituximab
- Golcadomide Dose 2 + Rituximab (Experimental)
  Interventions: Drug: Golcadomide; Drug: Rituximab

INTERVENTIONS:
Drug: Golcadomide — Specified dose on specified days
  Other Names: CC-99282; BMS-986369
  Arms: Golcadomide Dose 1 + Rituximab; Golcadomide Dose 2 + Rituximab
Drug: Rituximab — Specified dose on specified days
  Other Names: Mabthera
Drug: Cyclophosphamide — Specified dose on specified days
  Other Names: Endoxan
  Arms: Rituximab + Chemotherapy
Drug: Doxorubicin — Specified dose on specified days
  Other Names: Caelyx; pegylated liposomal doxorubicin; PLD
  Arms: Rituximab + Chemotherapy
Drug: Vincristine — Specified dose on specified days
  Arms: Rituximab + Chemotherapy
Drug: Prednisone — Specified dose on specified days
  Arms: Rituximab + Chemotherapy
Drug: Bendamustine — Specified dose on specified days
  Arms: Rituximab + Chemotherapy

SUMMARY:
The purpose of this study is to assess the efficacy and safety of golcadomide in combination with rituximab in participants with newly diagnosed advanced stage Follicular Lymphoma (FL).

ELIGIBILITY:
Inclusion Criteria

* Participant has histologically confirmed Grade 1, 2 or 3a follicular lymphoma (FL) or classic FL. Formalin-fixed paraffin embedded (FFPE) archival tissue from 1 year prior to screening is allowed. If more than 1 year has passed, then a fresh biopsy must be obtained to confirm the diagnosis.
* Have no prior systemic treatment for follicular lymphoma. Prior radiation therapy or surgery for previously diagnosed stage I disease is acceptable.
* Stage II to IV disease.
* Deemed to need treatment by treating investigator. Reasons for treatment can include, but are not limited to, the following:.

  i) Bulky disease defined as:.

A. A nodal or extra nodal (except spleen) mass > 7cm in its greater diameter or, involvement of at least 3 nodal or extra nodal sites (each with a diameter greater than >3 cm).

ii) Presence of at least one of the following B symptoms:.

A. Fever (>38°C) of unclear etiology.

B. Night sweats.

C. Weight loss greater than 10% within the prior 6 months.

iii) Splenomegaly with inferior margin below the umbilical line.

iv) Any one of the following cytopenia due to lymphoma:.

A. Platelets <100,000 cells/mm3 (100 x 109/L).

B. Absolute neutrophil count (ANC) < 1,000 cells/mm3 (1.0 x 109/L).

C. Hemoglobin < 10g/dL (6.25 mmol/L).

v) Pleural or peritoneal serous effusion (irrespective of cell content).

vi) Any compressive syndrome (for example, but not restricted to ureteral, orbital, gastrointestinal).

Exclusion Criteria

* Clinical evidence of transformed lymphoma by investigator assessment.
* Follicular Large Cell as per WHO 5th classification or Grade 3b follicular lymphoma as per WHO 4th classification.
* Participant has any significant medical condition, active infection, laboratory abnormality, or psychiatric illness that would prevent the participation in the study.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-11-23 (Estimated); Study Completion 2028-11-27 (Estimated)

PRIMARY OUTCOMES:
Number of participants who achieve complete metabolic response (CMR) as assessed by Lugano criteria 2014 | Up to approximately 12 months from participant randomization
  Golcadomide + Rituximab arms only

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) criteria, v.5.0 | Up to 28 days after last dose
Number of participants with Treatment-emergent AEs (TEAEs) as assessed by the NCI CTCAE criteria, v.5.0 | Up to 28 days after last dose
Best Overall Response (OR) | Up to approximately 12 months from participant randomization
  Defined as achieving CMR or partial metabolic response (PMR) based on Lugano criteria 2014
Duration of Response (DoR) | Up to approximately 3 years after randomization of the last participant
  Defined as time from first confirmed response (Complete Response (CR) or Partial Response (PR)) to disease progression, start of new anti-lymphoma therapy, or death
Complete Response at 30 months (CR30) | At approximately 30 months from randomization
  Defined as achieving CR based on Lugano criteria at 30 months from randomization
Complete Metabolic Response at 6 months from the randomization (CMR6) | At approximately 6 months from randomization
  Defined as achieving CMR based on Lugano criteria 2014 at 6 months from randomization
Complete Metabolic Response at 12 months from the randomization (CMR12) | At approximately 12 months from randomization
  Defined as achieving CMR based on Lugano criteria 2014 at 12 months from randomization
Progression Free Survival (PFS) | Up to approximately 3 years from randomization of last participant
  Defined as time from date of randomization to first occurrence of disease progression or death from any cause
Overall Survival (OS) | Up to approximately 3 years from randomization of last participant
  Defined as time from date of randomization to death from any cause
Number of participants who achieve CMR as assessed by Lugano criteria 2014 | Up to approximately 6 months from randomization
  Rituximab + Chemotherapy arm only

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (56):
- United States (18):
  - Local Institution - 0152, Birmingham, Alabama
  - Local Institution - 0055, Anchorage, Alaska
  - Local Institution - 0180, Phoenix, Arizona
  - Local Institution - 0190, Tucson, Arizona
  - Local Institution - 0035, San Francisco, California
  - Local Institution - 0022, Washington D.C., District of Columbia
  - Local Institution - 0209, Fort Myers, Florida
  - Local Institution - 0005, Jacksonville, Florida
  - Local Institution - 0210, St. Petersburg, Florida
  - Local Institution - 0026, Tampa, Florida
  - Local Institution - 0208, West Palm Beach, Florida
  - Local Institution - 0019, Westwood, Kansas
  - Local Institution - 0031, Rochester, Minnesota
  - Local Institution - 0111, Henderson, Nevada
  - Local Institution - 0183, Hackensack, New Jersey
  - Local Institution - 0052, Salt Lake City, Utah
  - Local Institution - 0201, Norfolk, Virginia
  - Local Institution - 0202, Seattle, Washington
- Australia (3):
  - Local Institution - 0046, Liverpool, New South Wales
  - Local Institution - 0070, South Brisbane, Queensland
  - Local Institution - 0181, Traralgon, Victoria
- Brazil (4):
  - Local Institution - 0061, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0060, Rio de Janeiro
  - Local Institution - 0058, São Paulo
  - Local Institution - 0056, São Paulo
- Canada (2):
  - Local Institution - 0064, Toronto, Ontario
  - Local Institution - 0205, Chicoutimi, Quebec
- Chile (2):
  - Local Institution - 0049, Santiago, Santiago Metropolitan
  - Local Institution - 0050, Santiago, Santiago Metropolitan
- France (4):
  - Local Institution - 0101, Saint-Cloud, Hauts-de-Seine
  - Local Institution - 0103, Lille, Nord
  - Local Institution - 0121, Poitiers, Vienne
  - Local Institution - 0118, Paris
- Germany (3):
  - Local Institution - 0197, Regensburg, Bavaria
  - Local Institution - 0188, Chemnitz, Saxony
  - Local Institution - 0189, Dresden
- Italy (4):
  - Local Institution - 0198, Rome, Lazio
  - Local Institution - 0179, Rozzano, Milano
  - Local Institution - 0076, Bologna
  - Local Institution - 0075, Napoli
- Poland (3):
  - Local Institution - 0187, Skórzewo, Greater Poland Voivodeship
  - Local Institution - 0186, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Local Institution - 0185, Warsaw, Masovian Voivodeship
- South Korea (3):
  - Local Institution - 0100, Busan, Pusan-Kwangyǒkshi
  - Local Institution - 0085, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0086, Seoul, Seoul-teukbyeolsi [Seoul]
- Spain (3):
  - Local Institution - 0196, Palma, Balears [Baleares]
  - Local Institution - 0192, Valencia, Valenciana, Comunitat
  - Local Institution - 0191, Madrid
- Taiwan (3):
  - Local Institution - 0094, Kaohsiung City
  - Local Institution - 0092, Kaohsiung City
  - Local Institution - 0123, Taipei
- United Kingdom (4):
  - Local Institution - 0175, Southampton, Hampshire
  - Local Institution - 0112, Canterbury, Kent
  - Local Institution - 0115, Edinburgh, Midlothian
  - Local Institution - 0105, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06425302.html